CLINICAL TRIAL: NCT02829242
Title: Near Infrared Spectroscopy for Determination of Tissue Oxygenation in Patients Undergoing Robotic Assisted Laparoscopic Surgery in the Trendelenburg Position - A Feasibility Study
Brief Title: Near Infrared Spectroscopy in Patients Undergoing Robotic Assisted Laparoscopic Surgery in the Trendelenburg Position
Status: Terminated | Type: Observational
Why Stopped: No sufficient patient recruitment
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Kabon, MD, Medical University of Vienna
Other Study IDs: NIRS_RALS
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Nontraumatic Compartment Syndrome of Leg
Keywords: Near Infrared Spectroscopy; Somatic Saturation; Well Leg Compartment Syndrome; Robotic Assisted Laparoscopic Surgery; Trendelenburg Position

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prostatic Surgery: Patient scheduled for a robotic assisted laparoscopic prostatic surgery.
  Interventions: Device: NIRS Monitoring (SenSmart Monitor)
- Colorectal Surgery: Patient scheduled for a robotic assisted laparoscopic colorectal surgery.
  Interventions: Device: NIRS Monitoring (SenSmart Monitor)

INTERVENTIONS:
Device: NIRS Monitoring (SenSmart Monitor)

SUMMARY:
Some robotic endoscopic surgeries require a steep Trendelenburg position and a carbon dioxide pneumoperitoneum. This minimally invasive approach has the advantages of less postoperative pain, shorter hospital stay and faster recovery. After prolonged operative time in a Trendelenburg position rare but significant complications are a cerebral oedema or a well leg compartment syndrome.

Well leg compartment syndrome results from inadequate perfusion in the lower limbs and the perfusion pressure is decreased proportionally to the lower extremity elevation. The condition can lead to release of intracellular proteins and myoglobinuria, hyperpotassaemia and metabolic acidosis followed by cell necrosis. The risk for tissue damage increases after 4 hours in a Trendelenburg position.

If not promptly diagnosed and treated, a compartment syndrome has devastating complications like permanent dysfunction, limb loss, renal failure or even death.

There are no specific guidelines for diagnosis and for the timing of surgical decompression. Fasciotomy is a clinical decision. There is no universal agreement at which compartment pressure irreversible muscle damage occurs.

The only objective diagnostic tool available is currently to measure the intramuscular pressure, however this is invasive, painful and may yield unreliable results. An intracompartment pressure of 0- 10mm Hg is the normal range.

Near Infrared Spectroscopy (NIRS) monitors are validated and approved to measure cerebral and somatic tissue oxygenation below the sensors and may help detecting promptly a compartment syndrome.

Therefore, the investigators designed the present study to detect a change in the tissue oxygenation in the lower legs during robotic assisted, laparoscopic surgery in the Trendelenburg position.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for robotic assisted laparoscopic surgery in a Trendelenburg position

Exclusion Criteria:

* Preexisting moderate neurological disease
* Moderate cerebrovascular disease
* Coronary disease with angina pectoris (CCS ≥ 1)
* Peripheral arterial disease II (with intermittent claudicatio)
* Cardiac insufficiency (NYHA >2)
* Tumour in pharynx, larynx or oesophagus, an aneurysm of the thoracic aorta

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Department of Surgery
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-07; Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Tissue oxygenation in the lower limbs during surgery in the Trendelenburg position. | during the operation
  Change over time in tissue oxygenation in the lower limbs during surgery in the Trendelenburg position.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No